CLINICAL TRIAL: NCT06844942
Title: Vessel Imaging Using Optical Coherence Tomography for Plaque Morphology and Vessel Fractional Flow Reserve
Acronym: VISION-FFR
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Mariusz Tomaniak, MD, PhD, Assoc. Prof., Medical University of Warsaw
Other Study IDs: VISION-FFR
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Tomography, Optical Coherence; 3D-angio-based FFR
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing coronary angiogram in chronic coronary syndrome with intermediate stenosis.: Patients undergoing coronary angiogram due to chronic coronary syndrome with intermediate grade coronary stenosis.
  Interventions: Diagnostic Test: vessel Fractional Flow Reserve

INTERVENTIONS:
Diagnostic Test: vessel Fractional Flow Reserve — Optical coherence tomography and vessel fractional flow reserve evaluation of coronary arteries with intermediate to severe stenosis.

SUMMARY:
The aim of this prospective, investigator-initiated study is to evaluate the diagnostic accuracy and correlations between mopphometric indices: luminal and qualitative parameters assessed by optical coherence tomography (OCT) including minimal lumen area, plaque type, presence of thin cap fibroatheroma and a functional index - angiography based vessel fractional flow reserve (vFFR) among patients with chronic coronary syndrome identified with intermediate grade coronary stenosis.

DETAILED DESCRIPTION:
This is a prospective, single center, non-randomized, single-arm, investigator-initiated study evaluating diagnostic accuracy and correlations between morphometric indices: luminal and qualitative parameters evaluated by optical coherence tomography (OCT) including minimal lumen area, plaque stratification into fibrotic, calcific, lipidic plaque, or thin cap fibroatheroma and a functional index - angiography based vessel fractional flow reserve (vFFR) among patients with chronic coronary syndrome identified with intermediate grade coronary stenosis.

The additional objectives encompass assessing the influence of age, sex, diabetes mellitus, renal dysfunction on the relationship between vFFR results and morphometric indices of intermediate coronary stenosis.

We hypothesized that in patients with intermediate grade coronary stenosis in chronic coronary syndrome a positive correlation exists between vFFR and the morphometric parameters associated with coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chronic coronary syndrome defined as presence of chest pain ranked 2-3 in the Canadian Cardiovascular Society classification or positive ischemia test (exercise test, single photon emission tomography (SPECT)
* Intermediate grade coronary stenosis of 40-80% assessed visually in coronary angiography and OCT examination The patient is willing to participate in the study and has provided a written informed consent

Exclusion Criteria:

* Acute coronary syndrome
* Proximal left main lesion
* Ostial right coronary artery lesion
* Bypass of the assessed vessel
* Contraindications for adenosine administration
* Hemodynamic instability
* Heart insufficiency in New York Heart Association (NYHA) class IV scale
* Acute renal insufficiency
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiogram due to chronic coronary syndrome with intermediate grade coronary stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between vessel fractional flow reserve (FFR) and minimal lumen area within the coronary stenosis | 0 days
  Correlation between vessel fractional flow reserve (FFR) and minimal lumen area within the coronary stenosis

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 36 months
  Major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department and Clinic of Cardiology, Medical University of Warsaw, Warsaw, Mazowieckie Voivodenship, Poland

IPD SHARING:
Plan to Share IPD: No